CLINICAL TRIAL: NCT03444571
Title: PRO-DIAG: Improved Diagnosis of Prosthetic Joint Infections
Acronym: PRO-DIAG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Yijuan Xu, Post Doc, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: PRO-DIAG; 27751 (Other Grant/Funding Number: Det Obelske Familiefond)
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Prosthesis-Related Infections
MeSH Terms: conditions — Prosthesis-Related Infections | interventions — Reoperation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- DNA based diagnosis (Experimental)
  Interventions: Procedure: revision surgery

INTERVENTIONS:
Procedure: revision surgery — If DNA based diagnosis detects infection, standard revision surgery will be conducted
  Arms: DNA based diagnosis

SUMMARY:
Implantation of joint prostheses is currently the second largest diagnosis-related group in the Danish health service, and in view of the demographic development and spread of lifestyle diseases, this type of intervention is expected to continue to increase.

Unfortunately, 5% of patients experience significant discomforts and complications. The second most frequent and serious complication is infection. While the established laboratory analyses (culture of tissue biopsies) are good at diagnosing acute infections, they are not satisfactory to diagnose a large group of patients especially with chronic infections. This can lead to prolonged diagnosing time and even to wrong diagnosis.

Several studies have shown that analyses of prosthetic parts and the use of molecular biological methods for detecting infecting microorganisms can significantly improve diagnostics accuracy.

The purpose of this project is primarily to demonstrate that analyses of bacterial specific DNA (16S rRNA genes) can confirm or rule out infection as fast (or faster) as cultivation methods. Rapid clarification can promote targeted treatment and in order to demonstrate this, the trial is conducted as a randomized study. .

ELIGIBILITY:
Inclusion Criteria:

* revision of hip platelets (THA) or knee replacement (TKA) on indication of likely infection

Exclusion Criteria:

* surgery within the last 4 months. The same applies to patients with short history of illness, pronounced acute symptoms and systemic response (reducing the likelihood of biofilm infection).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-02-16 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Improved diagnostic accuracy | 6 months post surgery
  DNA based method can detect patients with hidden chronic infections more often than culture

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic surgery, Aalborg, Northern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided